CLINICAL TRIAL: NCT04460508
Title: Efficacy and Safety of Mecapegfilgrastim(PEG-G-CSF) for Prophylaxis of Chemotherapy-induced Neutropenia in Patients With Lymphoma: a Randomized, Open-label, Active-controlled Trial
Brief Title: Mecapegfilgrastim(PEG-G-CSF) for Prophylaxis of Chemotherapy-induced Neutropenia in Patients With Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ou Bai, MD/PHD, Professor, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: mecapegfilgrastim-lym-2020-1
Record Dates: First submitted 2020-06-28; First posted 2020-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Chemotherapy-induced Neutropenia; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegylated granulocyte colony-stimulating factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mecapegfilgrastim (Experimental): Patients were administered pegylated rhG-CSF 6mg once at the 3rd day of every chemotherapy cycle.
  Interventions: Drug: Pegylated rhG-CSF
- rhG-CSF (Active Comparator): Patients were administered pegylated rhG-CSF 6 ug/kg/day from the 3rd day of every chemotherapy cycle.
  Interventions: Drug: rhG-CSF

INTERVENTIONS:
Drug: Pegylated rhG-CSF — Pegylated rhG-CSF:6mg
  Arms: Mecapegfilgrastim
Drug: rhG-CSF — rhG-CSF:5ug/kg/d
  Arms: rhG-CSF

SUMMARY:
Neutropenia is one of the most frequent adverse effects of chemotherapy, and the main factor to limit the dosage and the continuation of chemotherapy.A newly pegylated rhG-CSF was independently developed by JIANGSU HENGRUI Medicine Co., Ltd, China. Phase 1a, 1b and phase 2 trials have shown that pegylated rhG-CSF has decreased renal clearance, increased plasma half-life, and prolonged efficacy in compare with ﬁlgrastim.

This study is to evaluate efficacy and safety in chemotherapy-induced neutropenia of once-per-cycle Mecapegfilgrastim Injection(PEG-G-CSF) and daily G-CSF in Patients with lymphoma patients.

DETAILED DESCRIPTION:
This is a randomized, controlled study. A total of 170 lymphoma patients who are eligible are planned to randomized assigned into two groups to receive mecapegfilgrastim fixed dose of 6 mg or filgrastim 5 µg/kg/day during chemotherapy.

The primary endpoint is the duration of grade ≥3 neutropenia in cycle 1. The secondary endpoints include incidence of grade ≥3 neutropenia and febrile neutropenia (FN) in cycle 1-4, The pharmacoeconomics and safety profile are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years;
2. Patients with primary malignant lymphoma confirmed by histopathology or immunomolecular biology and requiring treatment with multi-cycle high-intensity chemotherapy regimen;
3. ECOG performance status ≤ 1;
4. ANC ≥1.5×109/L, PLT≥80×109 /L, Hb≥ 75g/L, WBC ≥3.0×109/L;
5. Subjects with pregnancy ability must agree to use reliable contraceptive measures from screening to 1 year after treatment;
6. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedul.

Exclusion Criteria:

1. Lymphoma central involvement;
2. Recipients of hematopoietic stem cell transplantation or organ transplantation;
3. Currently conducting clinical trials of other drugs;
4. There is an uncontrollable infection with body temperature ≥38℃;
5. liver function examination: total bilirubin (TBIL., alanine aminotransferase (ALT. and ascetic aminotransferase (AST. were all 2.5 times the upper limit of the normal value of >; if they were caused by liver metastasis, the upper limit of the normal value of > was 5 times;Renal function test: serum creatinine (Cr. >2 times the upper limit of normal value
6. Patients with serious chronic diseases of heart, kidney, liver and other important organs;
7. Patients with severe uncontrolled diabetes;
8. Pregnant or lactating female patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-03-20 (Estimated)

PRIMARY OUTCOMES:
Duration of grade ≥3 neutropenia in cycle 1 | 21 days
  Duration of subjects developing ANC lower than 1.0 × 109/L

SECONDARY OUTCOMES:
Incidence of grade ≥3 neutropenia in cycle 1-4 | 84 days
  Proportion of subjects developing ANC lower than 1.0 × 109/L from cycle 1 to cycle 4
Incidenc of febrile neutropenia (FN) in cycle 1-4 | 84 days
  Febrile neutropenia means the ANC count is less than 1,000/mm3 and body temperature is more than 38.5 degrees celsius from cycle 1 to cycle 4
Incidence of adverse events (AEs) | 84 days
  Analysis of adverse events (AEs) are based on treatment-related AEs (trAEs) according to the Common Terminology Criteria for Adverse Events, version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China